CLINICAL TRIAL: NCT06682507
Title: High Quality Evidence of Guangzhou Lupus Nephritis Cohort (HOPE Cohort)
Acronym: HOPE
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wei Chen, Director of Department of Nephrology, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: FirstSunYetSen2016-215
Record Dates: First submitted 2024-11-01; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Lupus Nephritis (LN)
Keywords: lupus; lupus nephritis; outcomes; end stage kidney disease
MeSH Terms: conditions — Lupus Nephritis; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Renal tissue from renal biopsy, urine, serum, DNA, PBMC, stool.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention: Observational Cohort

SUMMARY:
The goal of this observational study is to learn about the long-term renal and patient's survival of lupus nephritis (LN) patients in China. The main question it aims to answer is:

Does the renal and patient's survival improved in the long term period? Participants who had renal biopsy proven lupus nephritis in one hospital will be followed up.

DETAILED DESCRIPTION:
Patients from 1996-2016 were retrospective enrolled and patients starting from 2017 were prespective enrolled

ELIGIBILITY:
Inclusion Criteria:

Patients who had biopsy proven lupus nephritis in The First Affiliated Hospital of Sun Yat-sen University

Exclusion Criteria:

* less than 14 years old
* refused to give written consent

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had biopsy proven lupus nephritis in The First Affiliated Hospital of Sun Yat-sen University
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 1996-01-01 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with end stage renal disease | From data of enrollment until the data of first documented end stage renal disease, assessed up to 50 years
  End stage renal disease

SECONDARY OUTCOMES:
Rate of patient's mortality | From data of enrollment until the data of death, assessed up to 50 years
  death

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, MD PHD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data may contain privacy.